CLINICAL TRIAL: NCT01099202
Title: A Randomized Study of Procrit Versus No Procrit in Patients With Acute Lymphocytic Leukemia, Lymphoblastic Lymphoma, or Burkitt's Undergoing Induction/Consolidation Chemotherapy
Brief Title: Procrit Versus No Procrit in Acute Lymphocytic Leukemia, Lymphoblastic Lymphoma, or Burkitt's Undergoing Induction/Consolidation Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID02-591
Record Dates: First submitted 2010-04-05; First posted 2010-04-06 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: Procrit; Acute Lymphocytic Leukemia; Lymphoblastic Lymphoma; Burkitt's; Chemotherapy; Hyper-CVAD; augmented BFM; Epoetin alfa; Epogen; Erythropoietin
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Epoetin Alfa; Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Procrit (Experimental): Starting dose 40,000 units subcutaneously once a week with chemotherapy.
  Interventions: Drug: Procrit (epoetin alfa)
- No Procrit (No Intervention): No intervention.

INTERVENTIONS:
Drug: Procrit (epoetin alfa) — Starting dose 40,000 Units subcutaneously once a week during your regularly scheduled chemotherapy for up to 6 courses of chemotherapy (around 5 months).
  Other Names: epoetin alfa; Epogen; Erythropoietin
  Arms: Procrit

SUMMARY:
The goal of this clinical research study is to learn if Procrit (epoetin alfa) will decrease the need for blood transfusions in patients with Acute Lymphocytic Leukemia (ALL), Lymphoblastic Lymphoma (LL), or Burkitt's who are receiving chemotherapy. Another goal is to study the remission rates in patients with cancer who have received treatment with epoetin alfa.

DETAILED DESCRIPTION:
Epoetin alfa is a medication that helps the body make more red blood cells.

Before treatment you will have a complete physical exam. You will have around 1 tablespoon of blood drawn for blood tests (these tests are in addition to the routine blood tests you will have as part of your standard of care). Women who are able to have children must have a negative blood pregnancy test.

You will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Patients in the first group will be given epoetin alfa once a week at the time chemotherapy is started. Patients in the other group will not receive epoetin alfa, but will undergo the same laboratory exams and quality of life evaluations as the group of patients who were given epoetin alfa.

Patients in both groups will receive transfusions if their hemoglobin drops below a certain level or it the doctor feels it is necessary. These transfusions are considered to be standard of care. You will be asked to keep a diary listing the dates of all transfusions you receive.

If you are assigned to receive epoetin alfa, you will be given epoetin alfa once a week during your regularly scheduled chemotherapy. You will receive treatment with epoetin alfa for up to 6 courses of chemotherapy (usually around 5 months, but may be longer). Epoetin alfa will be given to you as an injection under the skin. Once a week, you will have around 1 tablespoon of blood drawn to check the level of hemoglobin in your blood. If your hemoglobin rises above a certain level, treatment with epoetin alfa may be temporarily stopped until your hemoglobin level decreases.

Patients in both groups will continue to receive chemotherapy during this study as scheduled. During chemotherapy, you will have around 1 tablespoon of blood drawn every 1-2 weeks for routine blood tests (as part of your standard of care for treatment of cancer).

If you agree to the optional procedures, you will continue receiving epoetin alfa even if your hemoglobin levels show that you are not responding to epoetin alfa treatment. However, if you do not choose to take part in the optional procedures and you are not responding to epoetin alfa treatment, you will be taken off the study.

If you experience any intolerable side effects that are a result of epoetin alfa or your disease gets worse, you will be taken off the study.

This is an investigational study. Epoetin alfa is FDA approved and commercially available. Around 164 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of ALL, LL, or Burkitt's receiving induction chemotherapy with Hyper-CVAD, any variant of Hyper-CVAD or augmented BFM at MD Anderson Cancer Center.
2. Patients must be enrolled on the study + / - (plus or minus) 14 days from the start of induction chemotherapy.
3. Patients with relapsed ALL, LL, or Burkitt's are eligible, but must have had a remission duration of 1 year or longer.

Exclusion Criteria:

1. Hemoglobin greater than or equal to 10 g/dL.
2. Patients with prior treatment with epoetin alfa or any investigational forms of erythropoietin within the previous 3 months.
3. Patients with known hypersensitivity to mammalian-cell derived products or to human albumin.
4. Uncontrolled hypertension
5. History of thrombotic vascular event.
6. Pregnant or lactating women.
7. Anemia due to factors other than cancer, deficiencies of B12, folate, or iron (only with concurrent treatment of these deficiencies).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2003-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 3/11/2003 - 5/25/2011; all patients were registered at The University of Texas M.D. Anderson Cancer Center.
Period: Overall Study
Arm/Group | Procrit | No Procrit
Started | 55 | 54
Completed | 55 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Procrit | No Procrit | Total
Number analyzed (Participants) | 55 | 54 | 109
Age Continuous [Median (Full Range); unit: years] | 39 [18 to 76] | 42 [15 to 84] | 41 [15 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 33 | 24 | 57
Region of Enrollment [Number; unit: participants]
  United States | 55 | 54 | 109

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of RBC Units Transfused During Initial 5 Months of Treatment
Description: Total number of packed red blood cell (PRBCs) units transfused to participant beginning at fifth week, up until 5-months compared between the evaluable study group subsets.
Time Frame: 5 weeks to 5 Months
Population: Transfusion data was available in 79 of the 81 (98%) evaluable patients who completed the treatment/observation period.
Measure: Mean (Standard Deviation); unit: PRBC Units
Groups:
- Procrit: Procrit starting dose 40,000 Units subcutaneously once a week with chemotherapy.
Arm/Group | Procrit | No Procrit
Number analyzed (Participants) | 41 | 38
PRBC Units | 10.63 (6.29) | 13.11 (5.18)

2. Primary Outcome: Number of PRBC Transfusions During Initial 5 Months of Treatment
Description: Total number of all packed red blood cells (PRBCs) transfusions (events) given to a participant throughout the 6 courses of chemotherapy treatment, collected and reported by participant from fifth week beginning baseline to 5 months.
Time Frame: 5 weeks to 5 Months
Population: Transfusion data was available in 79 of the 81 (98%) evaluable patients who completed the treatment/observation period.
Measure: Mean (Standard Deviation); unit: transfusions
Arm/Group | Procrit | No Procrit
Number analyzed (Participants) | 41 | 38
transfusions | 6.22 (3.87) | 7.44 (3.28)

ADVERSE EVENTS:
Time Frame: 8 years, 2 months
Arm/Group | Procrit | No Procrit
Serious Adverse Events (participants affected / at risk) | 8/55 | 6/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procrit (N=55) | No Procrit (N=54)
Deep Vein Thrombosis (Cardiac disorders) | 3 (3) | 2 (2)
Infection (Infections and infestations) | 5 (5) | 2 (2)
Seizures (Nervous system disorders) | 1 (1) | 2 (2)
Pulmonary Embolism (Cardiac disorders) | 1 (1) | 0 (0)
Stroke (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No